CLINICAL TRIAL: NCT00245570
Title: A Double-Blind, Randomized Multicenter, 3-Period, Crossover Study to Evaluate the Effects of a Single Dose of Montelukast Compared With Placebo and Salmeterol on Exercise-Induced Bronchoconstriction
Brief Title: Montelukast Compared With Placebo and Salmeterol in Exercise-Induced Bronchoconstriction (0476-316)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 0476-316; MK0476-316; 2005_043
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Results first posted 2010-05-27 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Asthma, Exercise-Induced
MeSH Terms: conditions — Asthma, Exercise-Induced | interventions — montelukast; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): Montelukast - Salmeterol - Placebo
  Interventions: Drug: Comparator: Montelukast; Drug: Comparator: Salmeterol; Drug: Comparator: Placebo (montelukast); Drug: Comparator: Placebo (salmeterol)
- 2 (Experimental): Montelukast - Placebo - Salmeterol
  Interventions: Drug: Comparator: Montelukast; Drug: Comparator: Salmeterol; Drug: Comparator: Placebo (montelukast); Drug: Comparator: Placebo (salmeterol)
- 3 (Experimental): Salmeterol - Montelukast - Placebo
  Interventions: Drug: Comparator: Montelukast; Drug: Comparator: Salmeterol; Drug: Comparator: Placebo (montelukast); Drug: Comparator: Placebo (salmeterol)
- 4 (Experimental): Salmeterol - Placebo - Montelukast
  Interventions: Drug: Comparator: Montelukast; Drug: Comparator: Salmeterol; Drug: Comparator: Placebo (montelukast); Drug: Comparator: Placebo (salmeterol)
- 5 (Experimental): Placebo - Montelukast - Salmeterol
  Interventions: Drug: Comparator: Montelukast; Drug: Comparator: Salmeterol; Drug: Comparator: Placebo (montelukast); Drug: Comparator: Placebo (salmeterol)
- 6 (Experimental): Placebo - Salmeterol - Montelukast
  Interventions: Drug: Comparator: Montelukast; Drug: Comparator: Salmeterol; Drug: Comparator: Placebo (montelukast); Drug: Comparator: Placebo (salmeterol)

INTERVENTIONS:
Drug: Comparator: Montelukast — 1 dose montelukast 10 mg tablet given orally in one of three treatment periods
Drug: Comparator: Salmeterol — 1 dose of 50 ug salmeterol given by inhalation in one of three treatment periods
Drug: Comparator: Placebo (montelukast) — 1 dose matching-image placebo to montelukast tablet in two of three treatment periods
Drug: Comparator: Placebo (salmeterol) — 1 dose matching-image placebo of salmeterol 50 ug inhalation in two of three treatment periods

SUMMARY:
To determine the effect of an approved medication being studied in support of a new approach in the prevention of exercise-induced asthma (a worsening of asthma caused by exercise, also known as exercise-induced bronchospasm), in patients who have a history of worsening asthma after exercise.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed exercise-induced bronchospasm

Exclusion Criteria:

* Patient is, other than asthma, not in good, stable health. The Primary Investigator will evaluate whether there are other reasons why the patient may not participate.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2005-12; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Philip G, Pearlman DS, Villaran C, Legrand C, Loeys T, Langdon RB, Reiss TF. Single-dose montelukast or salmeterol as protection against exercise-induced bronchoconstriction. Chest. 2007 Sep;132(3):875-83. doi: 10.1378/chest.07-0550. Epub 2007 Jun 15. PMID 17573489

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized at 5 sites (4 in the US and 1 in Peru).
  Primary therapy period: December 2005 to August 2006
Pre-assignment Details: Patients who required excluded medications, or did not meet FEV1 criteria during the prestudy period were excluded from randomization.
Groups:
- Montelukast/ Salmeterol/Placebo: During Period I (placebo run-in), all patients received a single witnessed dose of montelukast matching-image placebo oral tablet followed immediately by salmeterol matching-image placebo inhalation powder. During Period II, patients received a single witnessed dose of montelukast 10-mg oral tablet and salmeterol matching-image placebo inhalation powder.
  Washout 1 (Washout between Periods II and III) 3- to 7-day washout between Periods II and III.
  During Period III, patients received a single witnessed dose of montelukast matching-image placebo oral tablet followed immediately by salmeterol 50-μg inhalation powder.
  Washout 2 (Washout between Periods III and IV) 3- to 7-day washout between Periods III and IV.
  During Period IV, patients received a single witnessed dose of montelukast matching-image placebo oral tablet followed immediately by salmeterol matching-image placebo inhalation powder.
- Montelukast/ Placebo/ Salmeterol: During Period I (placebo run-in), all patients received a single witnessed dose of montelukast matching-image placebo oral tablet followed immediately by salmeterol matching-image placebo inhalation powder. During Period II, patients received a single witnessed dose of montelukast 10-mg oral tablet and salmeterol matching-image placebo inhalation powder.
  Washout 1 (Washout between Periods II and III) 3- to 7-day washout between Periods II and III.
  During Period III, patients received a single witnessed dose of montelukast matching-image placebo oral tablet followed immediately by salmeterol matching-image placebo inhalation powder.
  Washout 2 (Washout between Periods III and IV) 3- to 7-day washout between Periods III and IV.
  During Period IV, patients received a single witnessed dose of montelukast matching-image placebo oral tablet followed immediately by salmeterol 50-μg inhalation powder.
- Salmeterol / Montelukast/ Placebo: During Period I (placebo run-in), all patients received a single witnessed dose of montelukast matching-image placebo oral tablet followed immediately by salmeterol matching-image placebo inhalation powder. During Period II, patients received a single witnessed dose of montelukast matching-image placebo oral tablet followed immediately by salmeterol 50-μg inhalation powder.
  Washout 1 (Washout between Periods II and III) 3- to 7-day washout between Periods II and III.
  During Period III, patients received a single witnessed dose of montelukast 10-mg oral tablet and salmeterol matching-image placebo inhalation powder.
  Washout 2 (Washout between Periods III and IV) 3- to 7-day washout between Periods III and IV.
  During Period IV, patients received a single witnessed dose of montelukast matching-image placebo oral tablet followed immediately by salmeterol matching-image placebo inhalation powder.
- Salmeterol/ Placebo/ Montelukast: During Period I (placebo run-in), all patients received a single witnessed dose of montelukast matching-image placebo oral tablet followed immediately by salmeterol matching-image placebo inhalation powder. During Period II, patients received a single witnessed dose of montelukast matching-image placebo oral tablet followed immediately by salmeterol 50-μg inhalation powder.
  Washout 1 (Washout between Periods II and III) 3- to 7-day washout between Periods II and III.
  During Period III, patients received a single witnessed dose of montelukast matching-image placebo oral tablet followed immediately by salmeterol matching-image placebo inhalation powder.
  Washout 2 (Washout between Periods III and IV) 3- to 7-day washout between Periods III and IV.
  During Period IV, patients received a single witnessed dose of montelukast 10-mg oral tablet and salmeterol matching-image placebo inhalation powder.
- Placebo/ Montelukast/ Salmeterol: During Period I (placebo run-in), all patients received a single witnessed dose of montelukast matching-image placebo oral tablet followed immediately by salmeterol matching-image placebo inhalation powder. During Period II, patients received a single witnessed dose of montelukast matching-image placebo oral tablet followed immediately by salmeterol matching-image placebo
  inhalation powder.
  Washout 1 (Washout between Periods II and III) 3- to 7-day washout between Periods II and III.
  During Period III, patients received a single witnessed dose of montelukast 10-mg oral tablet and salmeterol matching-image placebo inhalation powder.
  Washout 2 (Washout between Periods III and IV) 3- to 7-day washout between Periods III and IV.
  During Period IV, patients received a single witnessed dose of montelukast matching-image placebo oral tablet followed immediately by salmeterol 50-μg inhalation powder.
- Placebo/ Salmeterol/ Montelukast: During Period I (placebo run-in), all patients received a single witnessed dose of montelukast matching-image placebo oral tablet followed immediately by salmeterol matching-image placebo inhalation powder. During Period II, patients received a single witnessed dose of montelukast matching-image placebo oral tablet followed immediately by salmeterol matching-image placebo inhalation powder.
  Washout 1 (Washout between Periods II and III) 3- to 7-day washout between Periods II and III.
  During Period III, patients received a single witnessed dose of montelukast matching-image placebo oral tablet followed immediately by salmeterol 50-μg inhalation powder.
  Washout 2 (Washout between Periods III and IV) 3- to 7-day washout between Periods III and IV.
  During Period IV, patients received a single witnessed dose of montelukast 10-mg oral tablet and salmeterol matching-image placebo inhalation powder.
Period: Treatment Period II
Arm/Group | Montelukast/ Salmeterol/Placebo | Montelukast/ Placebo/ Salmeterol | Salmeterol / Montelukast/ Placebo | Salmeterol/ Placebo/ Montelukast | Placebo/ Montelukast/ Salmeterol | Placebo/ Salmeterol/ Montelukast
Started | 7 | 8 | 8 | 8 | 8 | 8
Completed | 7 | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Between Periods II and III
Arm/Group | Montelukast/ Salmeterol/Placebo | Montelukast/ Placebo/ Salmeterol | Salmeterol / Montelukast/ Placebo | Salmeterol/ Placebo/ Montelukast | Placebo/ Montelukast/ Salmeterol | Placebo/ Salmeterol/ Montelukast
Started | 7 | 8 | 8 | 8 | 8 | 8
Completed | 7 | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period III
Arm/Group | Montelukast/ Salmeterol/Placebo | Montelukast/ Placebo/ Salmeterol | Salmeterol / Montelukast/ Placebo | Salmeterol/ Placebo/ Montelukast | Placebo/ Montelukast/ Salmeterol | Placebo/ Salmeterol/ Montelukast
Started | 7 | 8 | 8 | 8 | 8 | 8
Completed | 7 | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Between Periods III and IV
Arm/Group | Montelukast/ Salmeterol/Placebo | Montelukast/ Placebo/ Salmeterol | Salmeterol / Montelukast/ Placebo | Salmeterol/ Placebo/ Montelukast | Placebo/ Montelukast/ Salmeterol | Placebo/ Salmeterol/ Montelukast
Started | 7 | 8 (1 pt in the montelukast/placebo/salmeterol group discontinued during washout period 2 after placebo) | 8 | 8 | 8 | 8
Completed | 7 | 7 | 8 | 8 | 8 | 8
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Period: Treatment Period IV
Arm/Group | Montelukast/ Salmeterol/Placebo | Montelukast/ Placebo/ Salmeterol | Salmeterol / Montelukast/ Placebo | Salmeterol/ Placebo/ Montelukast | Placebo/ Montelukast/ Salmeterol | Placebo/ Salmeterol/ Montelukast
Started | 7 | 7 | 8 | 8 | 8 | 8
Completed | 7 | 7 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Population: All randomized patients
Arm/Group | Overall Study Population
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.0 (7.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 23
Need for β-agonist rescue medication following exercise challenge [Number; unit: participants]
  No | 31
  Yes | 16
Area under the FEV1 percent change from baseline time curve for 0-60 mins after exercise challenge [Mean (Standard Deviation); unit: % * minutes] | 957.46 (518.69)
Maximum percent fall in forced expiratory volume in 1 second (FEV1) post-exercise challenge [Mean (Standard Deviation); unit: Percent Change from Baseline] | 27.75 (6.26)
Time to recovery from maximal percent fall [Mean (Standard Deviation); unit: Minutes] — The duration between the time at which the maximum percent fall in FEV1 occurs and the time when FEV1 returns to within 5% of the preexercise baseline for the first time.
  Minutes | 55.03 (32.62)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Percent Fall in Forced Expiratory Volume in 1 Second (FEV1) After Exercise Challenge at 2 Hours Post-dose in Patients With Exercise-Induced Bronchoconstriction (EIB)
Description: In patients with EIB, the percent change from pre-exercise baseline FEV1 to the lowest FEV1 within 60 minutes after exercise challenge (2 hours post-dose). The FEV1 measurement obtained 5 minutes before the exercise challenge was the baseline, and was specific to each exercise challenge.
Time Frame: 0-60 minutes after the exercise challenge performed 2 hours after a single oral dose
Population: The primary efficacy analysis used the modified intention-to-treat (MITT) approach. Patients with data from only one period were not included in the analysis.
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline
Groups:
- Montelukast 10 mg: All Montelukast 10 mg patients from all Treatment Periods.
- Salmeterol 50-μg: All Salmeterol 50-μg patients from all Treatment Periods.
- Placebo: All Placebo patients from all Treatment Periods.
Arm/Group | Montelukast 10 mg | Salmeterol 50-μg | Placebo
Number analyzed (Participants) | 47 | 46 | 47
Percent Change from Baseline | 13.15 (10.28) | 10.46 (9.95) | 21.86 (13.44)

2. Secondary Outcome: Number of Patients Requiring β-Agonist Rescue Medication After Exercise Challenge at 2 Hours Postdose
Time Frame: 0-90 minutes after the exercise challenge performed at 2 hours postdose
Population: The secondary efficacy analysis used a modified intention-to-treat (MITT) approach. Patients with data from only one period were not included in the analysis.
Measure: Number; unit: Participants
Arm/Group | Montelukast 10 mg | Salmeterol 50-μg | Placebo
Number analyzed (Participants) | 47 | 46 | 47
Participants
  Patients Requiring Rescue Medication | 3 | 4 | 9
  Patients Not Requiring Rescue Medication | 44 | 42 | 38

3. Secondary Outcome: Number of Patients Requiring β-Agonist Rescue Medication After Exercise Challenge at 8.5 Hours Postdose
Time Frame: 0-90 minutes after the exercise challenge performed at 8.5 hours postdose
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Montelukast 10 mg | Salmeterol 50-μg | Placebo
Number analyzed (Participants) | 40 | 39 | 37
Participants
  Patients Requiring Rescue Medication | 0 | 0 | 4
  Patients Not Requiring Rescue Medication | 40 | 39 | 33

4. Secondary Outcome: Number of Patients Requiring β-Agonist Rescue Medication After Exercise Challenge at 24 Hours Postdose
Time Frame: 0-90 minutes after the exercise challenge performed at 24 hours postdose
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Montelukast 10 mg | Salmeterol 50-μg | Placebo
Number analyzed (Participants) | 46 | 46 | 46
Participants
  Patients Requiring Rescue Medication | 3 | 6 | 6
  Patients Not Requiring Rescue Medication | 43 | 40 | 40

5. Secondary Outcome: Maximum Percent Fall in FEV1 After Exercise Challenge at 8.5 Hours Post-dose in Patients With EIB
Description: In patients with EIB, the percent change from pre-exercise baseline FEV, to the lowest FEV1 within 60 minutes after exercise challenge (8.5 hours post-dose). The FEV1 measurement obtained 5 minutes before the exercise challenge was the baseline, and was specific to each exercise challenge.
Time Frame: 0-60 minutes after the exercise challenge performed 8.5 hours after a single oral dose
Population: The secondary efficacy analysis used the modified intention-to-treat (MITT) approach. Patients with data from only one period were not included in the analysis.
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline
Arm/Group | Montelukast 10 mg | Salmeterol 50-μg | Placebo
Number analyzed (Participants) | 40 | 39 | 37
Percent Change from Baseline | 11.60 (9.64) | 11.01 (7.56) | 16.65 (12.76)

6. Secondary Outcome: Maximum Percent Fall in FEV1 After Exercise Challenge at 24 Hours Post-dose in Patients With EIB
Description: In patients with EIB, the percent change from pre-exercise baseline FEV, to the lowest FEV1 within 60 minutes after exercise challenge (24 hours post-dose). The FEV1 measurement obtained 5 minutes before the exercise challenge was the baseline, and was specific to each exercise challenge.
Time Frame: 0-60 minutes after the exercise challenge performed 24 hours after a single oral dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline
Arm/Group | Montelukast 10 mg | Salmeterol 50-μg | Placebo
Number analyzed (Participants) | 46 | 46 | 46
Percent Change from Baseline | 10.09 (11.10) | 16.22 (13.09) | 13.64 (9.67)

7. Secondary Outcome: Area Under the Curve for FEV1 Percent Change From Preexercise Baseline During the 60 Minutes Following Exercise Challenge (AUC 0-60 Min) at 2 Hours Postdose
Description: The measure included only the area below the pre-exercise
  baseline
Time Frame: 0-60 minutes after the exercise challenge at 2 hours postdose
Population: The secondary efficacy analysis used a MITT approach. If a patient received β-agonist rescue medication during the 60 minutes following exercise challenge, then the last pre-rescue FEV1 measurement was carried forward to 60 minutes. Patients with data from only one period were not included in the analysis.
Measure: Mean (Standard Deviation); unit: Percent * minutes
Arm/Group | Montelukast 10 mg | Salmeterol 50-μg | Placebo
Number analyzed (Participants) | 47 | 46 | 47
Percent * minutes | 254.60 (241.17) | 293.05 (362.33) | 710.43 (529.91)

8. Secondary Outcome: Area Under the Curve for FEV1 Percent Change From Preexercise Baseline During the 60 Minutes Following Exercise Challenge (AUC 0-60 Min) at 8.5 Hours Postdose
Description: The measure included only the area below the pre-exercise baseline
Time Frame: 0-60 minutes after the exercise challenge at 8.5 hours postdose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent * minutes
Arm/Group | Montelukast 10 mg | Salmeterol 50-μg | Placebo
Number analyzed (Participants) | 40 | 39 | 37
Percent * minutes | 191.01 (166.24) | 276.26 (226.37) | 511.28 (566.30)

9. Secondary Outcome: Area Under the Curve for FEV1 Percent Change From Preexercise Baseline During the 60 Minutes Following Exercise Challenge (AUC 0-60 Min) at 24 Hours Postdose
Description: The measure included only the area below the pre-exercise baseline
Time Frame: 0-60 minutes after the exercise challenge at 24 hours postdose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent * minutes
Arm/Group | Montelukast 10 mg | Salmeterol 50-μg | Placebo
Number analyzed (Participants) | 46 | 46 | 46
Percent * minutes | 231.09 (413.73) | 554.93 (649.52) | 395.96 (464.92)

10. Secondary Outcome: Time to Recovery From Maximum Percentage Decrease in FEV1 After Exercise Challenge at 2 Hours Postdose
Description: The time to recovery from maximum percent fall is the duration between the time at which the maximum percent fall in FEV1 after exercise challenge occurs and the time when FEV1 returns to within 5% of the preexercise baseline for the first time.
Time Frame: Exercise challenge at 2 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Montelukast 10 mg | Salmeterol 50-μg | Placebo
Number analyzed (Participants) | 47 | 46 | 47
Minutes | 16.63 (23.72) | 17.58 (27.81) | 42.70 (34.26)

11. Secondary Outcome: Time to Recovery From Maximum Percentage Decrease in FEV1 After Exercise Challenge at 8.5 Hours Postdose
Description: as for outcome 10
Time Frame: Exercise challenge at 8.5 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Montelukast 10 mg | Salmeterol 50-μg | Placebo
Number analyzed (Participants) | 40 | 39 | 37
Minutes | 10.70 (13.38) | 13.82 (18.37) | 32.34 (34.57)

12. Secondary Outcome: Time to Recovery From Maximum Percentage Decrease in FEV1 After Exercise Challenge at 24 Hours Postdose
Description: as for outcome 10
Time Frame: Exercise challenge at 24 hours postdose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Montelukast 10 mg | Salmeterol 50-μg | Placebo
Number analyzed (Participants) | 46 | 46 | 46
Minutes | 11.04 (20.84) | 29.75 (33.50) | 23.31 (29.30)

ADVERSE EVENTS:
Time Frame: Periods II through IV and washout periods in between these treatment periods, and up to and including 14 days after the last dose of study therapy.
Description: Although a patient may have had two or more adverse experiences the patient is counted only once in a category. The same patient may appear in different categories.
Arm/Group | Montelukast/ Salmeterol/Placebo | Montelukast/ Placebo/ Salmeterol | Salmeterol / Montelukast/ Placebo | Salmeterol/ Placebo/ Montelukast | Placebo/ Montelukast/ Salmeterol | Placebo/ Salmeterol/ Montelukast
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.